CLINICAL TRIAL: NCT02430389
Title: Effect of Remifentanil Administration on Hemodynamic Stability During Placement of a Mayfield Head Fixation Device for Craniotomy
Brief Title: Effect of Remifentanil on Hemodynamic Stability During Placement of a Mayfield Head Fixation Device for Craniotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A priori hypothesis confirmed with interim analysis.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Laura Hemmer, Assistant Professor of Anesthesiology and Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00007835
Record Dates: First submitted 2015-04-25; First posted 2015-04-30 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Surgery
Keywords: hemodynamic stability; remifentanil
MeSH Terms: interventions — Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental): Intravenous bolus of 10 mL of remifentanil (0.7 mcg/kg based on ideal body weight) will be given ninety seconds before head pinning as well as an intravenous bolus of propofol (0.7 mg/kg).
  Interventions: Drug: Remifentanil
- Normal Saline (Placebo Comparator): Intravenous bolus of 10 mL normal saline from study syringe will be given ninety seconds before head pinning as well as an intravenous bolus of propofol (0.7 mg/kg).
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Remifentanil — Ninety seconds before pinning, an IV bolus of 10 mL of remifentanil (0.7 µg•kg-1 based on ideal body weight) will be administered from the study syringe and an IV bolus of propofol (0.7 mg•kg-1) will be administered
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Normal Saline — Ninety seconds before pinning, an IV bolus of 10 mL of normal saline will be administered from the study syringe and an IV bolus of propofol (0.7 mg•kg-1) will be administered
  Arms: Normal Saline

SUMMARY:
To identify a better method using a combination of routine anesthetic drugs to improve hemodynamic stability during Mayfield head pinning for craniotomy surgery.

DETAILED DESCRIPTION:
A randomized, placebo-controlled, double-blinded comparative effectiveness study to test hypothesis that addition of remifentanil bolus to a standard anesthetic drug regimen will better attenuate the hemodynamic response to the noxious stimulus of Mayfield head pin insertion than the standard anesthetic drug regimen.

ELIGIBILITY:
Inclusion Criteria:

* Adult non-pregnant patients
* undergoing general anesthesia for a craniotomy
* requiring a Mayfield head fixation device.

Exclusion Criteria:

* Patients under 18 years of age,
* non-English speaking,
* pregnancy,
* opioid tolerance,
* illegal drug use or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hemmer, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Cole CD, Gottfried ON, Gupta DK, Couldwell WT. Total intravenous anesthesia: advantages for intracranial surgery. Neurosurgery. 2007 Nov;61(5 Suppl 2):369-77; discussion 377-8. doi: 10.1227/01.neu.0000303996.74526.30. PMID 18091252
- [Background] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Background] Gazoni FM, Pouratian N, Nemergut EC. Effect of ropivacaine skull block on perioperative outcomes in patients with supratentorial brain tumors and comparison with remifentanil: a pilot study. J Neurosurg. 2008 Jul;109(1):44-9. doi: 10.3171/JNS/2008/109/7/0044. PMID 18590431
- [Background] Hans P, Brichant JF, Dewandre PY, Born JD, Lamy M. Effects of two calculated plasma sufentanil concentrations on the hemodynamic and bispectral index responses to Mayfield head holder application. J Neurosurg Anesthesiol. 1999 Apr;11(2):81-5. doi: 10.1097/00008506-199904000-00002. PMID 10213433
- [Background] Colley PS, Dunn R. Prevention of blood pressure response to skull-pin head holder by local anesthesia. Anesth Analg. 1979 May-Jun;58(3):241-3. No abstract available. PMID 572163
- [Background] Jamali S, Archer D, Ravussin P, Bonnafous M, David P, Ecoffey C. The effect of skull-pin insertion on cerebrospinal fluid pressure and cerebral perfusion pressure: influence of sufentanil and fentanyl. Anesth Analg. 1997 Jun;84(6):1292-6. doi: 10.1097/00000539-199706000-00022. PMID 9174309
- [Background] Coles JP, Leary TS, Monteiro JN, Brazier P, Summors A, Doyle P, Matta BF, Gupta AK. Propofol anesthesia for craniotomy: a double-blind comparison of remifentanil, alfentanil, and fentanyl. J Neurosurg Anesthesiol. 2000 Jan;12(1):15-20. doi: 10.1097/00008506-200001000-00004. PMID 10636615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Northwestern Memorial Hospital Ambulatory Surgery Unit or equivalent location where preoperative anesthesia evaluation occurring.
Groups:
- Remifentanil: Intravenous bolus of 10 mL of remifentanil (0.7 mcg/kg based on ideal body weight) will be given ninety seconds before head pinning as well as an intravenous bolus of propofol (0.7 mg/kg).
  Remifentanil: To determine if addition of remifentanil as an adjuvant with propofol will attenuate hemodynamic response to head pinning for the next ten minutes during and after pinning.
- Normal Saline: Intravenous bolus of 10 mL normal saline from study syringe will be given ninety seconds before head pinning as well as an intravenous bolus of propofol (0.7 mg/kg).
  Placebo
Period: Overall Study
Arm/Group | Remifentanil | Normal Saline
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Normal Saline | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.2) | 51.7 (4.8) | 56.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure After Head Fixation
Time Frame: Ten minute window after head fixation
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Remifentanil | Normal Saline
Number analyzed (Participants) | 10 | 10
mm Hg | 76 (8) | 83 (12)
Statistical Analysis 1: Comparison: Remifentanil vs Normal Saline; Test type: Superiority or Other; p = .0575, t-test, 2 sided

2. Secondary Outcome: Number of Patients Requiring Rescue Therapy for Hemodynamic Perturbations
Time Frame: 10 minute window after head fixation
Measure: Number; unit: participants
Arm/Group | Remifentanil | Normal Saline
Number analyzed (Participants) | 10 | 10
participants | 5 | 8
Statistical Analysis 1: Comparison: Remifentanil vs Normal Saline; Test type: Superiority or Other; p = .348, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 10 minutes post Mayfield head-pinning.
Description: In addition, patients were given contact information for study director if they had concerns of an adverse event or other concerns upon conclusion of study/recovery from anesthesia.
  Assessment of adverse reactions via chart review with need for rescue drug therapy.
Arm/Group | Remifentanil | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remifentanil (N=10) | Normal Saline (N=10)
hemodynamic perturbation (Cardiac disorders) | 5 (11) | 8 (31)

LIMITATIONS AND CAVEATS:
Study terminated early due to interim analysis with patients in placebo group having substantially higher systemic HTN requiring rescue meds compared to study drug group. Another limitation is difficulty defining baseline BP preoperatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes